CLINICAL TRIAL: NCT02159599
Title: An Open Label Randomized Clinical Trial, to Evaluate the Treatment With Darunavir/Ritonavir + Lamivudine Once Daily Versus Continuing With Darunavir/Ritonavir Once Daily + Tenofovir/Emtricitabine or Abacavir/Lamivudine in HIV Infected Subject With Suppressed Plasma Viremia
Brief Title: Study to Evaluate Darunavir/Ritonavir + Lamivudine Versus Continuing With Darunavir/Ritonavir + Tenofovir/Emtricitabine or Abacavir/Lamivudine in HIV Infected Subject
Acronym: DUAL
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Fundacion SEIMC-GESIDA (Other)
Collaborators: Janssen, LP (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: GESIDA 8014; 2014-000515-14 (EudraCT Number)
Record Dates: First submitted 2014-05-27; First posted 2014-06-10 (Estimated); Last update posted 2017-02-14 (Actual); Status verified 2016-06

CONDITIONS: HIV Infection
MeSH Terms: conditions — HIV Infections | interventions — Darunavir; Ritonavir; Lamivudine; Emtricitabine; Tenofovir; abacavir, lamivudine drug combination; Emtricitabine, Tenofovir Disoproxil Fumarate Drug Combination

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Darunavir/Ritonavir + 2 nucleos(t)idos (Active Comparator): Darunavir/Ritonavir ( (800mg/100mg) + Tenofovir/emtricitabine (300mg/200mg) or Abacavir/lamivudine (600 mg/300mg)
  Interventions: Drug: Darunavir/Ritonavir; Drug: Emtricitabine/tenofovir or abacavir/lamivudine
- Darunavir/ritonavir + Lamivudine (Experimental): Darunavir/Ritonavir (800mg7100mg) + lamivudine (300mg)
  Interventions: Drug: Darunavir/Ritonavir; Drug: Lamivudine

INTERVENTIONS:
Drug: Darunavir/Ritonavir — Darunavir/ritonavir (800/100 mg): QD (quaque die )
  Other Names: Prezista/Norvir
Drug: Lamivudine — Lamivudine (300mg) : QD
  Other Names: Epivir
  Arms: Darunavir/ritonavir + Lamivudine
Drug: Emtricitabine/tenofovir or abacavir/lamivudine — Emtricitabine/tenofovir (300/200 mg) or abacavir/lamivudine (600/300 mg): QD
  Other Names: Truvada or Kivexa
  Arms: Darunavir/Ritonavir + 2 nucleos(t)idos

SUMMARY:
This is an open label randomized clinial trial to evaluate the treatment with darunavir/ritonavir (800mg/100mg) plus lamivudine (300 mg) once daily versus continuing with darunavir/ritonavir (800mg/100mg) once daily plus tenofovir/emtricitabine (300mg/200mg) or abacavir/lamivudine (600mg/300mg) in HIV infected subject with suppressed plasma viremia.

ELIGIBILITY:
Inclusion Criteria:

1. Acceptance to participate in the study, signing the informed consent document before conducting any study procedures.
2. Patient with HIV infection older than 18 years.
3. Treatment with darunavir/ritonavir once a day and tenofovir/emtricitabine or abacavir/lamivudine during at least 4 weeks at the moment of the screening
4. Plasma HIV RNA levels below 50 copies / ml for at least 6 months (two separate measurements at least 6 months with viremia <50 copies / ml between both).
5. HbsAg negative

Exclusion Criteria:

1. Pregnant or breastfeeding woman
2. Evidence of Lamivudine resistance (any previous genotype with mutation M184V/I or K65R) and/or to darunavir (population genotype show any of the following mutations: V11I, V32I, L33F, I47V, I50V, I54L/M, G73S, T74P, L76V, I84V, L89V).
3. History of virology failure (two consecutive viral loads above 200 copies/ml) while the patient was receiving a regimen with lamivudine or emtricitabine, with the following exceptions:

   * Do not consider an exclusion criterion if the genotype performed at the time of failure does not demonstrate resistance to lamivudine and darunavir (see criteria 2).
   * Do not consider an exclusion criteria in the absence of genotype if after the episode turns to maintain a viral load <50 copies / ml with a treatment composed of lamivudine or emtricitabine + a nucleoside + a non-nucleoside.
4. History of abandonment of treatment including lamivudine or emtricitabine, with the following exception:

   - Viral load prior to abandonment was <50 copies / ml and subsequent reintroduction of the same treatment or another treatment consisting of lamivudine or emtricitabine + a nucleoside + a non-nucleoside returns to maintain viral load below 50 copies / ml .
5. Previous treatment with bitherapy or monotherapy with lamivudine or emtricitabine
6. Previous treatment with bitherapy or monotherapy with a regimen with a protease inhibitor that is terminated by viral rebound, when the absence of a genotypic resistance test available after viral rebound allow discard the resistance mutations either drug used.
7. The use of concomitant medication not permitted
8. Presence of active acute infection, including opportunist infection that a judge of investigator that can difficult the participation in the trial
9. Any laboratory results of the following: hemoglobin<8,0 g/dl; neutrophils <750 cells/µl; platelets <50.000 cell/µl; creatinine ≥ 1,5 ULN (upper limit of normal)
10. Any clinical or analytic event that, in the investigator judgment, condition the patient safety

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 249 (Actual)
Dates: Start 2014-07; Primary Completion 2016-04 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
Proportion of patients with undetectable viral load | week 48
  Undetectable viral load <50 copies/ml according to the FDA snapshot algorithm

SECONDARY OUTCOMES:
Proportion of patients with undetectable viral load | Week 24
  Undetectable viral load < 50 copies/ml according to the FDA snapshot algorithm
Proportion of patients with viral load < 200 copies/ml | week 48
  Proportion of patients with viral load < 200 copies/ml according to FDA snapshot algorithm
Proportion of patients who present viral load ≥ 50 copies /ml one time | From basal visit until week 48 visit
  Viral load ≥ 50 copies/ml
Proportion of patients who present viral load ≥ 50 copies /ml more tan two times | From basal visit until week 48 visit
  Viral load ≥ 50 copies /ml
Proportion of patients who maintained viral load < 50 copies/ml in all determinations | week 48
  Viral load < 50 copies/ml
Median of change cells CD4/µl count from basal to week 48 | week 48
  CD4/µl
Median of change in triglycerides , LDL-cholesterol, HDL-cholesterol and total cholesterol from basal to week 48 | week 48
Change in renal function | week 48
  Change in glomerular filtration
Change in proportion of patients with renal tubular dysfunction | week 48

OTHER OUTCOMES:
Proportion of genotypic resistance mutations | Week 48
  Mutations in patients viral failure
Change in proportion of genotypic resistance mutations | week 48

CONTACTS AND LOCATIONS:
Overall Officials: Jose R Arribas, MD, Study Director — Hospital Universitario La Paz; Federico Pulido, MD, Study Director — Hospital Universitario 12 de Octubre; Esteban Ribera, MD, Study Director — Hospital Vall d'Hebron
Locations (21):
- Spain (21):
  - Hospital Universitario de Bellvitge, L'Hospitalet de Llobregat, Barcelona
  - Hospital General Universitario de Alicante, Alicante
  - Hospital Universitario Germans Trias i Pujol, Badalona
  - Hospital Clinic, Barcelona
  - Hospital de La Santa Creu I Sant Pau, Barcelona
  - Hospital del Mar, Barcelona
  - Hospital Universitario Vall D'Hebron, Barcelona
  - Hospital Universitario Reina Sofía, Córdoba
  - Hospital Universitario Virgen de las Nieves, Granada
  - Complejo Hospitalario de Huelva, Huelva
  - Hospital 12 de Octubre, Madrid
  - Hospital Universitario Clínico San Carlos, Madrid
  - Hospital Universitario Fundación Alcorcón, Madrid
  - Hospital Universitario Gregorio Marañón, Madrid
  - Hospital universitario Infanta Leonor, Madrid
  - Hospital Universitario La Paz, Madrid
  - Hospital Universitario Príncipe de Asturias, Madrid
  - Hospital de Mataró, Mataró
  - Hospital Universitario Virgen de la Victoria, Málaga
  - Hospital Universitario Donostia, San Sebastián
  - Hospital Universitario Miguel Servet, Zaragoza

REFERENCES:
- [Derived] Pulido F, Ribera E, Lagarde M, Perez-Valero I, Palacios R, Iribarren JA, Payeras A, Domingo P, Sanz J, Cervero M, Curran A, Rodriguez-Gomez FJ, Tellez MJ, Ryan P, Barrufet P, Knobel H, Rivero A, Alejos B, Yllescas M, Arribas JR; DUAL-GESIDA-8014-RIS-EST45 Study Group. Dual Therapy With Darunavir and Ritonavir Plus Lamivudine vs Triple Therapy With Darunavir and Ritonavir Plus Tenofovir Disoproxil Fumarate and Emtricitabine or Abacavir and Lamivudine for Maintenance of Human Immunodeficiency Virus Type 1 Viral Suppression: Randomized, Open-Label, Noninferiority DUAL-GESIDA 8014-RIS-EST45 Trial. Clin Infect Dis. 2017 Nov 29;65(12):2112-2118. doi: 10.1093/cid/cix734. PMID 29020293